CLINICAL TRIAL: NCT03302351
Title: Comparing Dexmedetomidine, Ketamine and Dexmetedomidine-Ketamine Combination to Control Shivering During Regional Anaethesia
Brief Title: Dexmedetomidine, Ketamine and Dexmetedomidine-Ketamine Combination for Control of Shivering During Regional Anaethesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ghada Mohammed AboelFadl, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AMMH
Record Dates: First submitted 2017-09-26; First posted 2017-10-05 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Shivering
MeSH Terms: interventions — Dexmedetomidine; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dexmedetomidine (Experimental): 1st group will include 30 patients will receive intravenous dexmedetomidine 1 mcg/kg.
  Interventions: Drug: Dexmedetomidine
- Ketamine (Experimental): 2nd group will include 31 patients will receive intravenous ketamine 0.4 mg/kg.
  Interventions: Drug: ketamine
- Dexmetedomidine-Ketamine combination (Experimental): 3rd group will include 33 patients will receive combination between intravenous dexmedetomidine 0.5mcg/kg and low dose ketamine 0.25mg/kg.
  Interventions: Drug: Dexmetedomidine+Ketamine

INTERVENTIONS:
Drug: Dexmedetomidine — 30 patients will receive intravenous dexmedetomidine 1 mcg/kg.
  Other Names: precedex
  Arms: Dexmedetomidine
Drug: ketamine — 31 patients will receive intravenous ketamine 0.4 mg/kg.
  Other Names: katalar
  Arms: Ketamine
Drug: Dexmetedomidine+Ketamine — 33 patients will receive combination between intravenous dexmedetomidine 0.5mcg/kg + low dose ketamine 0.25mg/kg.
  Other Names: precedex+katalar
  Arms: Dexmetedomidine-Ketamine combination

SUMMARY:
Shivering is defined as an involuntary, repetitive activity of skeletal muscles. The incidence of shivering has been found to be quite high, approximately 40-50% in different studies. It can double or even triple oxygen consumption and carbon dioxide production. Shivering also increase intraocular and intracranial pressure, and may contribute to increased wound pain, delayed wound healing, and delayed discharge from post-anaesthetic care. Apart from being an uncomfortable experience, its deleterious effects deserve primary prevention and rapid control on occurence.

DETAILED DESCRIPTION:
Shivering is a physiological response to core hypothermia in an attempt to raise the metabolic heat production. The main causes of intra and postoperative shivering are heat loss, increased sympathetic tone, pain, and systemic release of pyrogens. Spinal anaesthesia significantly impairs the thermoregulation system by inhibiting tonic vasoconstriction, which plays a significant role in temperature regulation. It also causes a redistribution of core heat from the trunk (below the block level) to the peripheral tissues. These factors predispose patients to hypothermia and shivering.

The treatment of shivering includes both pharmacological and non-pharmacological methods. The non-pharmacological management is by external heating like the use of forced air warming, warming blankets, warmed fluids etc.

According to the results of meta-analysis, the most frequently reported pharmacological interventions include clonidine, pethidine, tramadol, nefopam, and ketamine. Unfortunately, no gold standard treatment is known for shivering as the administration of all the available drugs is associated with various adverse effects.

Dexmedetomidine, a congener of clonidine, is a highly selective adrenoceptor agonist. It has been used as a sedative agent and is known to reduce the shivering threshold. Few studies which have explored its anti-shivering potential have inferred that dexmedetomidine is an effective drug without any major adverse effect and provides good haemodynamic stability.

Ketamine has been tried to prevent shivering during anaesthesia with good results. Ketamine a competitive NMDA receptor antagonist has a role in thermoregulation at various levels. NMDA receptor modulates non-adrenergic and serotoninergic neurons in locus coeruleus. It is used as anti-shivering agent.

Shivering is a physiological response to core hypothermia in an attempt to raise the metabolic heat production. The main causes of intra and postoperative shivering are heat loss, increased sympathetic tone, pain, and systemic release of pyrogens. Spinal anaesthesia significantly impairs the thermoregulation system by inhibiting tonic vasoconstriction, which plays a significant role in temperature regulation. It also causes a redistribution of core heat from the trunk (below the block level) to the peripheral tissues. These factors predispose patients to hypothermia and shivering.

The treatment of shivering includes both pharmacological and non-pharmacological methods. The non-pharmacological management is by external heating like the use of forced air warming, warming blankets, warmed fluids etc.

According to the results of meta-analysis, the most frequently reported pharmacological interventions include clonidine, pethidine, tramadol, nefopam, and ketamine. Unfortunately, no gold standard treatment is known for shivering as the administration of all the available drugs is associated with various adverse effects.

Dexmedetomidine, a congener of clonidine, is a highly selective adrenoceptor agonist. It has been used as a sedative agent and is known to reduce the shivering threshold. Few studies which have explored its anti-shivering potential have inferred that dexmedetomidine is an effective drug without any major adverse effect and provides good haemodynamic stability.

Ketamine has been tried to prevent shivering during anaesthesia with good results. Ketamine a competitive NMDA receptor antagonist has a role in thermoregulation at various levels. NMDA receptor modulates non-adrenergic and serotoninergic neurons in locus coeruleus. It is used as anti-shivering agent.

ELIGIBILITY:
Inclusion Criteria:

* This study will include adults between 18 and 60 years of age undergo elective lower abdominal and lower limb surgery using spinal anaesthesia.
* ASA grade I - II

Exclusion Criteria:

* Patient refusal.
* Patients who have temperature over 37.3 or below 36 celsius degree.
* Known allergies to the study drugs.
* Contraindication to spinal anaesthesia as coagulopathy,
* patients with thyroid disease, Parkinson disease, dysautonomia, Raynaud syndrome, use of sedative-hypnotic agent or vasodilators.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
shivering score | 10 minutes
  p1(frequency of number)

CONTACTS AND LOCATIONS:
Locations (1):
- Ghada Mohammmad Aboalfadl, Asyut, Egypt

REFERENCES:
- [Background] Nikolic K, Popovic R. Conductometric determination of periciazine. Acta Pol Pharm. 1978;35(2):195-9. No abstract available. PMID 27062